CLINICAL TRIAL: NCT00253643
Title: Catechins and Omega-3 Fatty Acids Impact on Fatty Acid Synthase Activity in the Prostate: A Randomized Controlled Trial
Brief Title: Fish Oil and Green Tea Extract in Preventing Prostate Cancer in Patients Who Are at Risk for Developing Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jackie Shannon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000443617; P30CA069533 (NIH); OHSU-CI-CPC-04131-LX (Other: OHSU Knight Cancer Institute number); VAMC-04-0303/ M1016 (Other: Portland VA IRB number); DOD-W81XWH-04-1-0296 (Other Grant/Funding Number: Dept of Defense Award Number); OHSU-1117 (Other: OHSU IRB number); KPNW-NW-05SLIEB-01 (Other: Kaiser Permanente NW IRB number)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Precancerous Condition; Prostate Cancer
Keywords: prostate cancer; precancerous condition
MeSH Terms: conditions — Precancerous Conditions; Prostatic Neoplasms | interventions — polyphenon E; Fish Oils; Fatty Acids, Omega-3; Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (FO, GT catechin extract) (Experimental): Patients receive oral fish oil (FO) 3/day and oral green tea (GT) extract 2/day
  Interventions: Dietary Supplement: green tea catechin extract; Dietary Supplement: fish oil
- ArmII (FO placebo, GT catechin extract) (Experimental): Patients receive a fish oil (FO) placebo 3/day and oral green tea (GT) extract 2/day
  Interventions: Dietary Supplement: green tea catechin extract; Other: placebo
- Arm III (FO, GT placebo) (Experimental): Patients receive oral fish oil (FO) 3/day and a placebo mimicking green tea (GT) catechins 2/day
  Interventions: Dietary Supplement: fish oil; Other: placebo
- Arm IV (FO placebo, GT placebo) (Placebo Comparator): Patients receive a fish oil (FO) placebo mimicking fish oil 3/day and another placebo mimicking green tea (GT) catechins 2/day
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: green tea catechin extract — Given orally 2 times/day
  Other Names: Polyphenon E
  Arms: Arm I (FO, GT catechin extract); ArmII (FO placebo, GT catechin extract)
Dietary Supplement: fish oil — Given orally 3 times/day
  Other Names: omega-3 fatty acid, n-3 fatty acid, omega-3 polyunsaturated fatty acid, omega-3 PUFA
  Arms: Arm I (FO, GT catechin extract); Arm III (FO, GT placebo)
Other: placebo — Given olive oil placebo orally 3 times/day
  Other Names: PLCB, olive oil
  Arms: Arm III (FO, GT placebo); Arm IV (FO placebo, GT placebo)
Other: placebo — Given green tea placebo orally 2 times/day
  Other Names: PLCB
  Arms: Arm IV (FO placebo, GT placebo); ArmII (FO placebo, GT catechin extract)

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of fish oil and/or green tea may prevent prostate cancer.

PURPOSE: This randomized clinical trial is studying how well a fish oil and/or green tea supplement works in preventing prostate cancer in patients with prostatic intraepithelial neoplasia or who are at risk for developing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cancer preventing effects of fish oil supplementation and green tea extract use on markers of alteration in lipid metabolism in prostate tissue samples.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to age (under 65 vs 65 and over). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral fish oil three times daily and oral green tea extract twice daily.
* Arm II: Patients receive an oil placebo three times daily and oral green tea extract twice daily.
* Arm III: Patients receive oral fish oil three times daily and a placebo twice daily.
* Arm IV: Patients receive an oil placebo three times daily and another placebo twice daily.

Treatment in one of the above-listed arms continues for up to 20 weeks in the absence of disease progression or unacceptable toxicity.

All patients undergo a prostate biopsy on the last day of study treatment.

After completion of study treatment, patients receive a follow-up phone call at/around 30 days later.

PROJECTED ACCRUAL: A total of 144 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Clinician recommends repeat biopsy of the prostate ("Repeat" is defined as any recommended biopsy of the prostate subsequent to an earlier biopsy of the prostate)

EXCLUSION CRITERIA:

* Definitive invasive prostate cancer on initial biopsy
* Significant active medical illness that in the opinion of the clinician would preclude protocol treatment.
* History of ventricular tachycardia or ventricular fibrillation
* Subject reported use of fish oil (greater than 1 gram per day) or green tea supplement within 30 days before Day 1 of study treatment
* Subject reported use of fish oil ≤ 1 gram per day and unwilling to discontinue use for the duration of the trial
* Use of warfarin or need for therapeutic anticoagulation at time of biopsy or at anytime during the course of the trial.
* Subject reported allergy or sensitivity to fish oil, olive oil or green tea
* Subject reported history of hemophilia, van Willebrands disease or other bleeding disorder, except when the subject is evaluated by a hematologist who determines that fish oil supplementation is not contraindicated.
* Total bilirubin greater than institutional upper limit of normal
* Concurrent high risk study participation

Ages: 21 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-07; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon

REFERENCES:
- [Derived] Zhang Z, Garzotto M, Beer TM, Thuillier P, Lieberman S, Mori M, Stoller WA, Farris PE, Shannon J. Effects of omega-3 Fatty Acids and Catechins on Fatty Acid Synthase in the Prostate: A Randomized Controlled Trial. Nutr Cancer. 2016 Nov-Dec;68(8):1309-1319. doi: 10.1080/01635581.2016.1224365. Epub 2016 Sep 20. PMID 27646578

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Fish Oil, Green Tea Catechin Extract): Patients receive oral fish oil 3/day and oral green tea extract 2/day
  green tea catechin extract: Given orally 2 times/day
  fish oil: Given orally 3 times/day
  laboratory biomarker analysis: Correlative studies
  questionnaire administration: Ancillary studies
- Arm II (Fish Oil Placebo, Green Tea Catechin Extract): Patients receive an oil placebo 3/day and oral green tea extract 2/day
  green tea catechin extract: Given orally 2 times/day
  placebo: Given olive oil placebo orally 3 times/day
  laboratory biomarker analysis: Correlative studies
  questionnaire administration: Ancillary studies
- Arm III (Fish Oil, Green Tea Placebo): Patients receive oral fish oil 3/day and a placebo mimicking green tea catechins 2/day
  fish oil: Given orally 3 times/day
  placebo: Given green tea placebo orally 2 times/day
  laboratory biomarker analysis: Correlative studies
  questionnaire administration: Ancillary studies
- Arm IV (Fish Oil Placebo, Green Tea Placebo): Patients receive an oil placebo mimicking fish oil 3/day and another placebo mimicking green tea catechins 2/day
  placebo: Given olive oil placebo orally 3 times/day
  placebo: Given green tea placebo orally 2 times/day
  laboratory biomarker analysis: Correlative studies
  questionnaire administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Fish Oil, Green Tea Catechin Extract) | Arm II (Fish Oil Placebo, Green Tea Catechin Extract) | Arm III (Fish Oil, Green Tea Placebo) | Arm IV (Fish Oil Placebo, Green Tea Placebo)
Started | 14 | 15 | 29 | 31
Completed | 14 | 15 | 28 | 28
Not Completed | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Non-Compliance | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Fish Oil, Green Tea Catechin Extract): Patients receive oral fish oil 3/day and oral green tea extract 2/day
  green tea catechin extract: Given orally 2 times/day
  fish oil: Given orally 3 times/day
- Arm II (Fish Oil Placebo, Green Tea Catechin Extract): Patients receive an oil placebo 3/day and oral green tea extract 2/day
  green tea catechin extract: Given orally 2 times/day
  placebo: Given olive oil placebo orally 3 times/day
- Arm III (Fish Oil, Green Tea Placebo): Patients receive oral fish oil 3/day and a placebo mimicking green tea catechins 2/day
  fish oil: Given orally 3 times/day
  placebo: Given green tea placebo orally 2 times/day
- Arm IV (Fish Oil Placebo, Green Tea Placebo): Patients receive an oil placebo mimicking fish oil 3/day and another placebo mimicking green tea catechins 2/day
  placebo: Given olive oil placebo orally 3 times/day
  placebo: Given green tea placebo orally 2 times/day
- Total: Total of all reporting groups
Arm/Group | Arm I (Fish Oil, Green Tea Catechin Extract) | Arm II (Fish Oil Placebo, Green Tea Catechin Extract) | Arm III (Fish Oil, Green Tea Placebo) | Arm IV (Fish Oil Placebo, Green Tea Placebo) | Total
Number analyzed (Participants) | 14 | 15 | 28 | 28 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18 | 19 | 55
  >=65 years | 6 | 5 | 10 | 9 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 15 | 28 | 28 | 85
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 28 | 28 | 85
Diagnosis [Number; unit: participants]
  Benign | 9 | 11 | 16 | 21 | 57
  Prostate Cancer | 2 | 1 | 6 | 6 | 15
  Prostatic Intraepithelial Neoplasia (PIN) | 3 | 3 | 6 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Fatty Acid Synthase Expression by Immunohistochemistry at Pre- and Post-intervention (FAS Summary Score)
Description: Sections of paraffin-embedded prostate biopsy tissue were stained for fatty acid synthase (FAS) expression. The FAS Summary Score was calculated as the product of percent stained (1=0-25%, 2=25-50%, 3=51-75%, 4=76-100%) and stain intensity (0-3) by immunohistochemistry. The range of the product is 0-300.
Time Frame: Baseline (pre-intervention) and end of study (time to surgery for those with malignant findings or up to 8 weeks for those with benign biopsies, post-intervention)
Population: Number of participants for recruitment was based on power calculations. All participants consented and randomized were included in analyses. Analysis was intention to treat. No imputations for missing data were conducted.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm I: Fish oil, Green Tea catechin extract
- Arm II: Fish oil placebo, Green Tea catechin extract
- Arm III: Fish oil, Green Tea placebo
- Arm IV: Fish oil placebo, Green Tea placebo
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 14 | 15 | 28 | 28
units on a scale
  PRE data | 147 (98.6) | 158.8 (84.6) | 138.3 (63.8) | 102.3 (85.9)
  POST data | 140.7 (100.3) | 159.3 (75.5) | 145.2 (72.2) | 152.2 (80.9)
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Mixed effects model to assess the effect time (pre vs. post) and treatment (GTFO, GT, FO and Placebo) on FAS summary scores; Test type: Superiority or Other; p = 0.1521, Mixed Models Analysis — Utilized a priori threshold for statistical significance of 0.05

2. Primary Outcome: Cell Proliferation by Ki67-immunohistochemistry at Pre- and Post-intervention
Description: Cell Proliferation by Ki67 is calculated as the percent stained by immunohistochemistry. Ki-67 values were log-transformed because the original distribution was skewed. Analysis was done on log-base2 transformed values.
Time Frame: End of study
Population: as for outcome 1
Measure: Median (Full Range); unit: %age of cells & nuclei stained
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 14 | 15 | 28 | 28
%age of cells & nuclei stained | 18.5 [1 to 55] | 8 [2 to 52] | 10 [0 to 45] | 12 [1 to 50]
Statistical Analysis 1: Comparison: Arm I vs Arm II vs Arm III vs Arm IV; Mixed effects model to assess the effect of time (pre vs. post) and treatment (GTFO, GT, FO and Placebo) on Ki-67; Test type: Superiority or Other; p = 0.1573, Mixed Models Analysis — A priori threshold for statistical significance is 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every month the subject was on study via questionnaire over the phone. We conducted a 30-day follow-up phone call and utilized our adverse event questionnaire to capture this information at baseline as well.
Arm/Group | Arm I (Fish Oil, Green Tea Catechin Extract) | Arm II (Fish Oil Placebo, Green Tea Catechin Extract) | Arm III (Fish Oil, Green Tea Placebo) | Arm IV (Fish Oil Placebo, Green Tea Placebo)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 1/14 | 2/15 | 5/29 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Fish Oil, Green Tea Catechin Extract) (N=14) | Arm II (Fish Oil Placebo, Green Tea Catechin Extract) (N=15) | Arm III (Fish Oil, Green Tea Placebo) (N=29) | Arm IV (Fish Oil Placebo, Green Tea Placebo) (N=31)
Bloating (grade 2) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muscle Pain (grade 2) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Gas/Flatulence (grade 2) (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Burping (grade 2) (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea/Vomiting (grade 2) (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Bruising (grade 2) (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Headache (grade 2) (Nervous system disorders) | 0 | 0 | 2 | 1
Upset Stomach (grade 2) (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhea/ Loose Stool (grade 2) (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Heartburn (grade 2) (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes